CLINICAL TRIAL: NCT02883192
Title: The Effect of Preventive Use of Ondansetron on the Blood Pressure and Vasopressor Consumption in the Cesarean Section Under Spinal Anesthesia
Brief Title: The Effect of Preventive Use of Ondansetron in the Cesarean Section Under Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS.GAITINI, M.D., Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BnaiZionMC-16-LG-011
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Adverse Anesthesia Outcome
Keywords: Cesarean section; spinal anesthesia; hypotension; ondansetron
MeSH Terms: conditions — Hypotension | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ondansetron (Experimental): ondansetron
  Interventions: Drug: Ondansetron
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — Zofran 4 mg.
  Other Names: Zofran
  Arms: ondansetron
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Cesarean section is a frequent procedure in the obstetric surgery. The most widely used anesthesia technique for cesarean delivery is the spinal anesthesia The incidence of spinal anesthesia induced hypotension and bradycardia is high as 60% in the obstetric population. The aim of the study is to investigate the effect of the preventive use of Ondansetron on the prevention of hypotension

DETAILED DESCRIPTION:
Cesarean section is a frequent procedure in the obstetric surgery. The most widely used anesthesia technique for cesarean delivery is the spinal anesthesia, in our Institute over than 90% of the elective cesarean sections are under spinal anesthesia, however this kind of anesthesia frequently associated with, side effects that affect primarily the parturient and the fetal health. The incidence of spinal anesthesia induced hypotension and bradycardia is high as 60% in the obstetric population . Most authors agree that hypotension presents when the systolic blood pressure decrease under 90 mmHg, or when there is a reduction from baseline of more than 20-30 %. Augmentation of the intravascular volume with crystalloids and vasopressors is the cornerstone of the treatment of spinal anesthesia induced hypotension, the vasopressors usually used are the α and β receptors agonist ephedrine and the selective α agonist phenylephrine that, gain popularity in the last years, because it's more efficacy in maintaining the umbilical cord blood PH and the Apgar score of the neonates. However many studies showed that it was inefficient and no intervention reliably prevents hypotension after spinal anesthesia for cesarean section and, bradycardia can occur from shift in cardiac autonomic balance toward the parasympathetic system from activation of left ventricular mechanoreceptors after sudden decrease in left ventricle volume causing the Bezold Jarish Reflex (BJR). Animal studies suggest that 5-HT( serotonin) may play an important factor associated inducing the BJR and this effect can be blocked at the 5-HT3 receptor using the serotonin inhibitor Ondansetron, commonly used antiemetic . Despite the fact that Ondansetron was evaluated in the management of spinal anesthesia induced hypotension in large heterogeneity and small samples , the need for more investigation in big number of cesarean sections still needed.

The aim of the study is to investigate the effect of the preventive use of Ondansetron on the prevention of hypotension and the amount of vasopressor phenylephrine needed to control the hypotension after spinal anesthesia and the possible effect on the umbilical cord blood PH and the Apgar score in one minute after delivery.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesia (ASA) physical status I or II

Exclusion Criteria:

Preeclampsia Cardiovascular disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure measure in mmHg. | 40 minutes

SECONDARY OUTCOMES:
Vomiting measure in number scale | 40 minutes

CONTACTS AND LOCATIONS:
Overall Officials: mira koch, M.A., Study Chair — Bnai Zion Medical Center
Locations (1):
- Luis A Gaitini M.D., Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes